CLINICAL TRIAL: NCT00004039
Title: Phase II Trials of CHOP Chemotherapy and Interferon Alpha or Rituximab Anti-CD20 Monoclonal Antibody as Initial Treatment of Patients With Stage III and IV High-Risk Indolent B-Cell Lymphoma and Intermediate Grade B-Cell Lymphoma
Brief Title: Combination Chemotherapy Plus Interferon Alfa or Rituximab in Treating Patients With Stage III or Stage IV Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patient accruals
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Collaborators: Cancer Biotherapy Research Group (Other)
Responsible Party: Robert O. Dillman, MD, Hoag Memorial Hospital Presbyterian
Purpose: Treatment
Other Study IDs: CDR0000066762; CBRG-9807; NCI-V98-1494
Record Dates: First submitted 1999-12-10; First posted 2004-08-05 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Lymphoma
Keywords: Waldenstrom macroglobulinemia; stage II grade 3 follicular lymphoma; stage II adult diffuse small cleaved cell lymphoma; stage II adult diffuse mixed cell lymphoma; stage II adult diffuse large cell lymphoma; stage II adult immunoblastic large cell lymphoma; stage II adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult Burkitt lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell | interventions — Interferon-alpha; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: recombinant interferon alfa
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining interferon alfa or the monoclonal antibody rituximab with chemotherapy may kill more cancer cells.

PURPOSE: Phase II trial to compare the effectiveness of combination chemotherapy plus interferon alfa or rituximab in treating patients who have high risk stage III or stage IV lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) with either interferon alfa or rituximab in patients with stage III or IV high risk indolent or intermediate B-cell lymphoma. II. Determine the objective tumor response rate and duration of response for these regimens in these patients. III. Determine the failure free survival and overall survival for these patients on these regimens. IV. Compare the response rate and survival rate of these patients on these regimens to similar patients treated in published studies. V. Compare the toxicities of these regimens in these patients. VI. Determine the quality of life of these patients on these regimens.

OUTLINE: This is a multicenter study. Patients are assigned to one of two treatment arms: Arm I: Patients receive rituximab IV on day 0, and cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1, followed by oral prednisone on days 1-5. Arm II: Patients receive interferon alfa subcutaneously on days 22-26, and cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1, followed by oral prednisone on days 1-5. Treatment repeat every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline and prior to chemotherapy for each course. Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually for up to 10 years.

PROJECTED ACCRUAL: A total of 40-80 patients (20-40 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed high risk (stage III or IV) indolent or intermediate (stage II to IV) B-cell lymphoma Small cleaved cell lymphoma Waldenstrom's macroglobulinemia Follicular small cleaved cell or mixed cell Follicular large cell Diffuse Immunoblastic High risk is defined as: Increased LDH OR Increased beta-2-microglobulin OR B symptoms OR Bulky disease of greater than 7 cm in diameter OR Extranodal disease other than blood or bone marrow involvement OR Mantle zone histology At least 1 lymph node or visceral lesion at least 2 cm in diameter

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No active infection or other medical condition this is lifethreatening Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: No prior therapy for lymphoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1998-06; Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Cancer Biotherapy Research Group
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States